CLINICAL TRIAL: NCT05257889
Title: An Overview on Neonatal Seizures in Neonatal Intensive Care Unit of Assuit University Children's Hospital, a Cross Sectional Study
Brief Title: Neonatal Seizures in NICU of Assuit University Children's Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Salama, principal investigator, Assiut University
Other Study IDs: 17101539
Record Dates: First submitted 2022-02-07; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Neonatal Seizure
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — * CBC
  * Serum electrolytes (Serum Glucose, Serum Calcium , Serum Magnesium )
  * Liver function tests
  * Blood urea and Serum Creatinine
  * Blood gases
  * CSF only (in suspected cases of CNS infections)
  * Serum ammonia and lactate levels for neonates suspected to have inborn errors of metabolism (extended metabolic screen if possible)
  * TORCH screening
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neonatal seizures cases: Cases of neonatal seizures
  Interventions: Diagnostic Test: blood and CSF studies + neuroimaging studies
- seizure-free neonates: cases that are seizure free
  Interventions: Diagnostic Test: blood and CSF studies + neuroimaging studies

INTERVENTIONS:
Diagnostic Test: blood and CSF studies + neuroimaging studies — blood and CSF studies + neuroimaging studies

SUMMARY:
A cross sectional study on neonatal seizures in Assuit University Children's hospital NICU.

DETAILED DESCRIPTION:
An Overview on neonatal seizures in neonatal intensive care unit of Assuit University Children's hospital , a cross sectional study. The aim of this study is to evaluate the clinical seizures during the neonatal period and its prevalence

ELIGIBILITY:
Inclusion Criteria:

* ALL neonates (preterm and full-term infants) aged 0 to 28 days who are admitted to the neonatal intensive care unit of Assiut University Children's hospital during the period of the study will be included

Exclusion Criteria:

* Neonates with multiple congenital anomalies (other than CNS anomalies)

Ages: 1 Day to 1 Month | Sex: All
Age Groups: Child
Study Population: ALL neonates (preterm and full-term infants) aged 0 to 28 days who are admitted to the neonatal intensive care unit of Assiut University Children's hospital
Sampling Method: Non-Probability Sample
Enrollment: 554 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
prevalence of neonatal seizures among neonates admitted to Assiut University children's hospital | 1 year
  prevalence of neonatal seizures among neonates admitted to Assiut University children's hospital during period of study

SECONDARY OUTCOMES:
number of patients with controlled seizures during hospital admission period | 1 year
  Short term outcomes of clinical seizures (if seizures could be controlled during hospital admission period or not)

IPD SHARING:
Plan to Share IPD: Undecided